CLINICAL TRIAL: NCT05053256
Title: The Relationship Between Heart Function and Metabolism in Heart Failure With Preserved Ejection Fraction Patients
Brief Title: The Relationship Between Heart Function and Metabolism in HFpEF Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2021-08-29
Record Dates: First submitted 2021-08-30; First posted 2021-09-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF: Heart failure with preserved ejection fraction
- HFrEF: Heart failure with reduced ejection fraction

SUMMARY:
HFpEF has gradually become the most common form of heart failure. Studies have found that metabolic abnormalities and chronic inflammation ultimately lead to HFpEF by promoting heart remodeling. However, there are few relevant studies and the mechanism is still unclear.

DETAILED DESCRIPTION:
However, heart failure with preserved ejection fraction is difficult to diagnose and treat due to its unknown pathogenesis and poor prognosis. Ventricular diastolic dysfunction and retention of left ventricular ejection fraction are important pathological features of Heart failure with preserved ejection fraction. Currently, it is widely believed to be a clinical syndrome associated with old age, women, obesity, diabetes, hypertension, atrial fibrillation, coronary heart disease, atherosclerosis, etc. However, the specific mechanism of heart failure with preserved ejection fraction caused by the above-mentioned complications is unknown. In conclusion, the investigators intend to explore the pathogenesis of heart failure with preserved ejection fraction by observing the changes of heart and body metabolism in patients with heart failure with preserved ejection fraction, and provide a basis for the diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged ≥ 18 years old
* Patients diagnosed with HFpEF;

Diagnostic criteria including:

1. LVEF 50% or higher;
2. BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL;
3. Presence of symptoms and/or signs of heart failure;
4. At least one additional criteria: relevant structure heart disease or diastolic dysfunction

Exclusion Criteria:

* Severe liver failure;
* Other causes of shortness of breath, such as severe pulmonary disease or severe ● chronic obstructive pulmonary disease;
* Primary pulmonary hypertension.
* Severe left valvular heart disease.
* Long-term bedridden or unable to move autonomously
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | On admission
  The muscle mass of HFpEF patients, such as thigh muscle mass
Blood uric acid | On admission
  The blood uric acid of HFpEF patients
Body fat content | On admission
  The body fat content of HFpEF patients, such as fat percentage and visceral fat area.

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No